CLINICAL TRIAL: NCT03126786
Title: Randomized, Double Masked, Controlled Study Comparing the Safety and Efficacy of Suprachoroidal CLS-TA With Intravitreal Aflibercept Versus Aflibercept Alone in Subject With Diabetic Macular Edema
Brief Title: Suprachoroidal CLS-TA With Intravitreal Aflibercept Versus Aflibercept Alone in Subject With Diabetic Macular Edema
Acronym: TYBEE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS1004-201
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes Mellitus; Diabetic Retinopathy; Microneedle; Mircoinjection; Triamcinolone; Choroid; Choroid Injection; Aflibercept; Suprachoroidal; Triamcinolone acetonide
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — aflibercept; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Treatment will consist of IVT injection of Aflibercept followed by an SC injection of CLS-TA
  Interventions: Drug: IVT aflibercept; Drug: SC CLS-TA
- Control (Sham Comparator): Treatment will consist of IVT aflibercept injection followed by a sham SC procedure
  Interventions: Drug: IVT aflibercept; Drug: Sham SC

INTERVENTIONS:
Drug: IVT aflibercept — IVT aflibercept [2 mg/0.05 mL]
  Other Names: Eylea
Drug: Sham SC — sham SC
  Other Names: suprachoroidal sham
  Arms: Control
Drug: SC CLS-TA — CLS-TA [4 mg/100 μL] SC injection
  Other Names: Triamcinolone Acetonide
  Arms: Active

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of suprachoroidal CLS-TA used with intravitreal aflibercept in subjects with DME.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-masked, controlled, parallel-group study of 6 months duration in treatment-naïve subjects with DME. This study is projected to enroll approximately 60 subjects, randomly assigned 1:1 to one of two treatment groups.

The study design includes up to 8 clinic visits over approximately 24 weeks. Subjects will attend visits for Screening (Visit 1, Days -30 to 0); Randomization and Baseline (Visit 2, Day 0 before dosing); Dosing and Evaluation (Visit 2 after dosing to Visit 5, Day 0 through Week 12); As-needed (PRN) Dosing and Follow up (Visit 6 through Visit 7, Week 16 through Week 20), and End of Study (Visit 8, Week 24).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 or type 2 DM
* DME with central involvement (> 300 µm in the central subfield on spectral-domain optical coherence tomography [SD-OCT], in the study eye
* ETDRS BCVA score of ≥ 20 letters read and ≤ 70 letters read in the study eye
* Naïve to local pharmacologic treatment for DME in the study eye

Exclusion Criteria:

* IOP > 21 mmHg in the study eye at Visit 1 (Day -30 to -1); subjects are not excluded if IOP is <22 mmHg in the study eye with no more than 1 IOP lowering medication
* Any previous treatment in the study eye with an ocular corticosteroid implant
* Has significant media opacity precluding evaluation of retina and vitreous in the study eye.
* History of glaucoma or optic nerve head change consistent with glaucoma damage
* History of glaucoma surgery
* History of clinically significant IOP elevation in response to corticosteroid treatment ("steroid responder")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical
Locations (29):
- United States (29):
  - Retinal Consultants of Arizona and Retinal Research Institute, Phoenix, Arizona
  - Retina Centers, PC, Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Medical Group Clinical Research, Beverly Hills, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - Retina Institute of California, Palm Desert, California
  - Retina Consultants San Diego, Poway, California
  - MedEye Associates, Miami, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Emory Eye Center, Augusta, Georgia
  - Marietta Eye Clinic, Marietta, Georgia
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina and Vitrous Associates of Kentucky, Lexington, Kentucky
  - The Johns Hopkins Wilmer Eye Institute, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Associates of NJ, Teaneck, New Jersey
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Oregon Retina Institute, Medford, Oregon
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates-Arlington, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Treatment will consist of IVT injection of Aflibercept followed by an SC injection of CLS-TA
  IVT aflibercept: IVT aflibercept [2 mg (0.05 mL)]
  SC CLS-TA: SC CLS-TA [40 mg/mL]
- Control: Treatment will consist of IVT aflibercept injection followed by a sham SC procedure
  IVT aflibercept: IVT aflibercept [2 mg (0.05 mL)]
  Sham SC: sham SC
Period: Overall Study
Arm/Group | Active | Control
Started | 36 | 35
Completed | 30 | 33
Not Completed | 6 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Safety population included all randomly assigned subjects who were administered at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of subject, in years, relative to the date of the Screening Visit.
  years | 59.8 (10.16) | 59.2 (12.89) | 59.5 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Biological gender of the subject.
  Participants
    Female | 10 | 11 | 21
    Male | 26 | 24 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnic background as reported by the subject.
  Participants
    Hispanic or Latino | 12 | 9 | 21
    Not Hispanic or Latino | 24 | 26 | 50
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race as reported by the subject.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 2 | 5
    White | 31 | 32 | 63
    More than one race | 0 | 1 | 1
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Region of participation by the subject.
  participants
    United States | 36 | 35 | 71
Best corrected visual acuity [Mean (Standard Deviation); unit: letters] — Best corrected visual acuity letter score following refraction and Early Treatment Diabetic Retinopathy Study protocol.
  letters | 57.1 (13.00) | 58.1 (11.33) | 57.6 (12.13)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity Letter Score
Description: Best corrected visual acuity (BCVA) refers to the measurement of the best possible vision that can be achieved following refraction or correction. BCVA was assessed following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol and was measured in the number of letters read correctly on an ETDRS eye chart. An increase from the pre-treatment state in BCVA of 15 letters or more represents a clinically meaningful improvement.
Time Frame: Baseline, 6 months
Population: The Intent-to-treat population included all randomized subjects who received at least 1 study treatment
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Active | Control
Number analyzed (Participants) | 36 | 35
letters | 11.4 (1.63) | 13.8 (1.59)
Statistical Analysis 1: Comparison: Active vs Control; The primary efficacy analysis comparing ACTIVE with CONTROL on the mean change from baseline (Visit 2, Day 0) BCVA at Week 12 was be performed using a Mixed Model for Repeated Measurements (MMRM). This model included treatment (ACTIVE or CONTROL), visit (Visit 3 (Week 4), Visit 4 (Week 8), and Visit 5 (Week 12), Visit 6 (Week 16), Visit 7 (Week 20) and Visit 8 (Week 24), and the 2-way interactions of treatment and visit, and the BCVA baseline included as the covariate; Test type: Superiority — The sample size was determined such that the difference in visual acuity between the ACTIVE treatment group and CONTROL treatment group could be estimated within +/- five ETDRS letters. Week 24 data from the Eylea prescribing information was used to estimate a pooled standard deviation of 9.17 letters. With 28 subjects per arm, a two-sided 90% confidence interval with a distance from the mean difference to the limits (half of interval width) will be less than 5 letters; p = 0.288, Mixed model for repeat measures — There was a single primary outcome tested at a single primary endpoint, therefore no adjustments for multiple comparisons were performed. The primary endpoint was assess with a 2-sided alpha level of 0.100; The covariance structure was assumed to be unstructured; Mean Difference (Final Values) = -2.4, 90% CI 2-sided [-6.2 to 1.4], Standard Error of Mean 2.28 — Estimated Value calculated as Active minus Control

2. Secondary Outcome: Mean Change From Baseline in Central Subfield Thickness
Description: Central subfield thickness (CST) is a diagnostic measurement used in identifying the presence of edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT). A masked reading center graded the SD-OCT digital images. A negative change from baseline value represents a reduction in macular edema.
Time Frame: Baseline, 6 months
Population: The Intent-to-treat population included all randomized subjects who received at least 1 study treatment
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | Active | Control
Number analyzed (Participants) | 36 | 35
microns | -212.1 (13.83) | -178.6 (13.61)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 24 weeks of follow-up.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 2/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/36 | 4/35
Other Adverse Events (participants affected / at risk) | 10/36 | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=36) | Control (N=35)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=36) | Control (N=35)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 3 (3) | 4 (4)
Intraocular pressure increased (Eye disorders) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (5)
Retinal exudates (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institutions and Investigators participating in this study shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical, Inc.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT03126786/Prot_SAP_000.pdf